# Self-Image Research Study – Informed Consent (E) Union College

**Researchers:** D. Catherine Walker, Ph.D. and undergraduate psychology research assistants, Emily Ehrlich and Meichai Chen, both affiliated with Union College in Schenectady, NY.

**Research Description:** This self image research study aims to test the impact of undergraduate women's response to guided mirror exposure and texts that prompt them to focus on gratitude.

**Human Subject Involvement:** Research participants will be asked to partake in a three-week long program with a one-month and a four month follow-up assessment. All assessment sessions will include answering questions about topics such as mood, self-image, attitudes about the self, self-esteem, and typical self-care behaviors (e.g., eating and physical activity). Participants will be asked to respond to gratitude journaling text prompts three days a week during the three week-long program. Participants will also be asked to participate in weekly mirror exposure exercises. During the mirror exposure exercise, participants will be asked to direct their attention to specific body parts and may be asked to think about or describe those body parts based on their features. Each weekly session in the lab will likely last approximately an hour for the three weeks of participation, as well as the follow up assessments. We ask that participants do not participate in a Union College Body Project Workshop until after the four month follow-up assessment.

**Risks and Discomforts of Participation:** Mirror exposures have been found to lead to temporary increases in psychological distress. However, that distress is short-lived (Shafran, Lee, Payne, & Fairburn, 2007). Ongoing research suggests that guided and unguided mirror exposure exercises lead to improvement in body image satisfaction among women with high body dissatisfaction (Díaz-Ferrer et al., 2017).

**Measures taken to minimize risks and discomfort:** The mirror exposure is not expected to have any long-term negative effects and may improve participants' body image satisfaction over time (Díaz-Ferrer et al., 2017). Participants are free to withdraw at any time without facing any penalty. Additionally, participants will be provided with a list of treatment resources.

**Expected benefits to subjects or to others:** Although we cannot promise you any direct benefit from your participation in this study, the knowledge gained may ultimately benefit other individuals who suffer from body image problems. In addition, you may also gain insight into some aspects of your own self-image and will be introduced to a potentially promising new intervention for self-image.

Confidentiality of records/data: All information obtained in this study is strictly confidential: the researcher promises not to divulge this information, unless disclosure is required by law. Information that you provide in the online questionnaires will be linked with a unique Participant Identification Number. Your name will only be linked to your Participant Identification Number on a password-protected computer file that can only be accessed by Dr. Walker. Research findings containing group data may be published; however, no personal information or individual questionnaire responses will be published. For text responses to gratitude questions, the research coordinator will be able to link your responses to your identity, but not to your survey questionnaires. However, the gratitude question text responses are not expected to be sensitive in content.

**Payment to subject for participation:** If participants choose to withdraw from the study, they will be compensated for the portions of the study that they have completed. The payment schedule is as follows: \$15 for the first week, \$10 for the second week, \$15 for the third week, \$15 for the 1 month follow up assessment, and

\$25 for the 4 month follow up assessment - for a **total of \$80** over the course of the study for participants who complete every session.

Contact information: If you have any questions about this study, please contact the Principal Investigator: D. Catherine Waker, Ph.D., Licensed Clinical Psychologist and Visiting Assistant Professor of Psychology at Union College, (518)-388-6538, walkerc@union.edu.

You will be offered a copy of this form to keep for your records.

**Your rights as a research participant:** Research at Union College involving human participants is carried out under the oversight of the Human Subjects Research Committee (HSRC). This research has been reviewed and approved by the HSRC. If you have any questions about your rights as a human research participant, more information can be found at the Office of Human Research Protections: https://www.hhs.gov/ohrp/

**Voluntary Nature of Participation:** Even after you agree to participate, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise are entitled. You can choose at any time not to answer a question, or not complete a portion of the research for any reason.

Withdrawal of subjects and data retention: Your participation in this project is voluntary. Even after you agree to participate in the research or sign the informed consent document, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise have been entitled. I will retain and analyze the information you have provided unless you request that your data be excluded from any analysis and/or destroyed.

Listed below are mental health resources in the even that you have concerns related to or are upset by any of the topics covered in this study.

- For emergency mental health services, call the Albany County Mental Health 24-hour Crisis Hotline at (518) 447-9650 or the Samaritan Hospital 24-Hour Crisis Line at (518) 274-4345.
- The National Eating Disorders Association helpline has a telephone and an online chat support: <a href="https://www.nationaleatingdisorders.org/help-support/contact-helpline">https://www.nationaleatingdisorders.org/help-support/contact-helpline</a>; Confidential helpline, Monday Thursday from 9:00 am 9:00 pm and Friday from 9:00 am 5:00 pm (EST): 1-800-931-2237
- The Union College Eppler-Wolff Counseling Center (for UAlbany students) located in the Wicker Wellness Center on Union College Campus; telephone: (518) 388-6161; email: uchealthcenter@union.edu
- The Psychological Services Center located at 299 Washington Avenue, Albany, NY 12206; telephone: (518) 442-4900. Offers therapy on a sliding scale based on income, with low rates for students.
- For intensive outpatient program (IOP) services for eating disorders: HPA/LiveWell located at 260 Washington Avenue Extension, Suite 101, Albany, NY 12203; telephone: (518) 218-1188 [Note: the P.I. in this study (DCW) is on staff at HPA/LiveWell as a clinical psychologist, so is aware of patients seen in the IOP. In this capacity, DCW is legally required to uphold patient confidentiality.]

4 641

,. .

| I have read, or been informed of, the information about thi | s study. I hereby consent to participate in the study. |
|---|---|
| Name: | |
| Signature: | Date: |

# Self-Image Research Study – Informed Consent (E) University at Albany

**Researchers:** D. Catherine Walker, Ph.D., Visiting Assistant Professor of Psychology at Union College and Volunteer Research Associate at University at Albany, State University of New York (Principal Investigator) and Drew A. Anderson, Ph.D., Associate Professor of Psychology at University at Albany, State University of New York, co-Principal Investigator.

**Research Description:** This self image research study aims to test the impact of undergraduate women's response to guided mirror exposure and texts that prompt them to focus on gratitude.

**Human Subject Involvement:** Research participants will be asked to partake in a three-week long program with a one-month and a four month follow-up assessment. All assessment sessions will include answering questions about topics such as mood, self-image, attitudes about the self, self-esteem, and typical self-care behaviors (e.g., eating and physical activity). Participants will be asked to respond to gratitude journaling text prompts three days a week during the three week-long program. Participants will also be asked to participate in weekly mirror exposure exercises. During the mirror exposure exercise, participants will be asked to direct their attention to specific body parts and may be asked to think about or describe those body parts based on their features. Each weekly session in the lab will likely last approximately an hour for the three weeks of participation, as well as the follow up assessments.

**Risks and Discomforts of Participation:** Mirror exposures have been found to lead to temporary increases in psychological distress. However, that distress is short-lived (Shafran, Lee, Payne, & Fairburn, 2007). Ongoing research suggests that guided and unguided mirror exposure exercises lead to improvement in body image satisfaction among women with high body dissatisfaction (Díaz-Ferrer et al., 2017).

**Measures taken to minimize risks and discomfort:** The mirror exposure is not expected to have any long-term negative effects and may improve participants' body image satisfaction over time (Díaz-Ferrer et al., 2017). Participants are free to withdraw at any time without facing any penalty. Additionally, participants will be provided with a list of treatment resources.

**Expected benefits to subjects or to others:** Although we cannot promise you any direct benefit from your participation in this study, the knowledge gained may ultimately benefit other individuals who suffer from body image problems. In addition, you may also gain insight into some aspects of your own self-image and will be introduced to a potentially promising new intervention for self-image.

Confidentiality of records/data: All information obtained in this study is strictly confidential: the researcher promises not to divulge this information, unless disclosure is required by law. Information that you provide in the online questionnaires will be linked with a unique Participant Identification Number. Your name will only be linked to your Participant Identification Number on a password-protected computer file that can only be accessed by Dr. Walker. Research findings containing group data may be published; however, no personal information or individual questionnaire responses will be published. For text responses to gratitude questions, the research coordinator will be able to link your responses to your identity, but not to your survey questionnaires. However, the gratitude question text responses are not expected to be sensitive in content.

**Payment to subject for participation:** If participants choose to withdraw from the study, they will be compensated for the portions of the study that they have completed. The payment schedule is as follows: \$15 for

the first week, \$10 for the second week, \$15 for the third week, \$15 for the 1 month follow up assessment, and \$25 for the 4 month follow up assessment - for a **total of \$80** over the course of the study for participants who complete every session.

Contact information: If you have any questions about this study, please contact the Principal Investigator: D. Catherine Waker, Ph.D., Licensed Clinical Psychologist and Visiting Assistant Professor of Psychology at Union College, (518)-388-6538, walkerc@union.edu.

You will be offered a copy of this form to keep for your records.

**Your rights as a research participant:** Research at Union College involving human participants is carried out under the oversight of the Human Subjects Research Committee (HSRC). This research has been reviewed and approved by the HSRC. If you have any questions about your rights as a human research participant, more information can be found at the Office of Human Research Protections: https://www.hhs.gov/ohrp/

**Voluntary Nature of Participation:** Even after you agree to participate, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise are entitled. You can choose at any time not to answer a question, or not complete a portion of the research for any reason.

Withdrawal of subjects and data retention: Your participation in this project is voluntary. Even after you agree to participate in the research or sign the informed consent document, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise have been entitled. I will retain and analyze the information you have provided unless you request that your data be excluded from any analysis and/or destroyed.

Listed below are mental health resources in the even that you have concerns related to or are upset by any of the topics covered in this study.

- For emergency mental health services, call the Albany County Mental Health 24-hour Crisis Hotline at (518) 447-9650 or the Samaritan Hospital 24-Hour Crisis Line at (518) 274-4345.
- The National Eating Disorders Association helpline has a telephone and an online chat support: <a href="https://www.nationaleatingdisorders.org/help-support/contact-helpline">https://www.nationaleatingdisorders.org/help-support/contact-helpline</a>; Confidential helpline, Monday Thursday from 9:00 am 9:00 pm and Friday from 9:00 am 5:00 pm (EST): 1-800-931-2237
- The University at Albany Counseling Center (for UAlbany students) located at 400 Patroon Creek Blvd Suite 104, Albany, NY 12206; email: consultation@albany.edu; telephone: (518) 442-5800.
- The Psychological Services Center located 299 Washington Avenue, Albany, NY 12206; telephone: (518) 442-4900.
- Counseling Care and Services located at 405 Vliet Boulevard, Cohoes, NY 12047; telephone: (518) 237-4263.
- For intensive outpatient program (IOP) services for eating disorders: HPA/LiveWell located at 260 Washington Avenue Extension, Suite 101, Albany, NY 12203; telephone: (518) 218-1188 [Note: the P.I. in this study (DCW) is on staff at HPA/LiveWell as a clinical psychologist, so is aware of patients seen in the IOP. In this capacity, DCW is legally required to uphold patient confidentiality.]

| Consent | 01 | the | par | ticij | pant | t: |
|---------|----|-----|-----|-------|------|----|
|---------|----|-----|-----|-------|------|----|

| Name: | - |
|------------|-------|
| Signature: | Date: |

I have read, or been informed of, the information about this study. I hereby consent to participate in the study.

# Self-Image Research Study – Informed Consent (C) Union College

**Researchers:** D. Catherine Walker, Ph.D., principal investigator, and undergraduate psychology research assistants, Emily Ehrlich and Meichai Chen, both affiliated with Union College in Schenectady, NY.

**Research Description:** This self image research study aims to test the impact of undergraduate women's response to guided mirror exposure and texts that prompt them to focus on gratitude.

**Human Subject Involvement:** Research participants will be asked to partake in a three-week long program with a one-month and a four month follow-up assessment. All assessment sessions will include answering questions about topics such as mood, self-image, attitudes about the self, self-esteem, and typical self-care behaviors (e.g., eating and physical activity). Each weekly session in the lab will likely last approximately a half hour for the three weeks of participation, as well as for each of the the follow-up assessments. We ask that participants do not participate in a Union College Body Project Workshop until after the four-month follow-up assessment.

**Risks and Discomforts of Participation:** We do not anticipate any risk in your participation. It is possible that you may become uncomfortable answering some of the questions. Please note that your participation in this study is completely **voluntary**.

Measures taken to minimize risks and discomfort: Participants will be provided with a list of local and national treatment resources.

**Expected benefits to subjects or to others:** Although we cannot promise you any direct benefit from your participation in this study, the knowledge gained may ultimately benefit other individuals who suffer from body image problems. In addition, you may also gain insight into some aspects of your own self-image and will be introduced to a potentially promising new intervention for self-image.

Confidentiality of records/data: All information obtained in this study is strictly confidential: the researcher promises not to divulge this information, unless disclosure is required by law. Information that you provide (in online questionnaires and via text) will be linked with a unique Participant Identification Number. Your name will only be linked to your Participant Identification Number on a password-protected computer file that can only be accessed by Dr. Walker. Research findings containing group data may be published; however, no personal information or individual questionnaire responses will be published.

**Payment to subject for participation:** If participants choose to withdraw from the study, they will be compensated for the portions of the study that they have completed. The payment schedule is as follows: \$10 for the first week, \$10 for the third week, \$15 for the 1 month follow up assessment, and \$25 for the 4 month follow up assessment - for a **total of \$60** over the course of the study for full participation.

Contact information: If you have any questions about this study, please contact the Principal Investigator: D. Catherine Waker, Ph.D., Licensed Clinical Psychologist and Visiting Assistant Professor of Psychology at Union College, (518)-388-6538, walkerc@union.edu. You will be offered a copy of this form to keep.

**Your rights as a research participant:** Research at Union College involving human participants is carried out under the oversight of the Human Subjects Research Committee (HSRC). This research has been reviewed and approved by the HSRC. If you have any questions about your rights as a human research participant, more information can be found at the Office of Human Research Protections: https://www.hhs.gov/ohrp/

**Voluntary Nature of Participation:** Even after you agree to participate, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise are entitled. You can choose at any time not to answer a question, or not complete a portion of the research for any reason.

Withdrawal of subjects and data retention: Your participation in this project is voluntary. Even after you agree to participate in the research or sign the informed consent document, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise have been entitled. I will retain and analyze the information you have provided unless you request that your data be excluded from any analysis and/or destroyed.

Listed below are mental health resources in the even that you have concerns related to or are upset by any of the topics covered in this study.

- For emergency mental health services, call the Albany County Mental Health 24-hour Crisis Hotline at (518) 447-9650 or the Samaritan Hospital 24-Hour Crisis Line at (518) 274-4345.
- The National Eating Disorders Association helpline has a telephone and an online chat support: <a href="https://www.nationaleatingdisorders.org/help-support/contact-helpline">https://www.nationaleatingdisorders.org/help-support/contact-helpline</a>; Confidential helpline, Monday Thursday from 9:00 am 9:00 pm and Friday from 9:00 am 5:00 pm (EST): 1-800-931-2237
- The Union College Eppler-Wolff Counseling Center (for UAlbany students) located in the Wicker Wellness Center on Union College Campus; telephone: (518) 388-6161; email: uchealthcenter@union.edu
- The Psychological Services Center located at 299 Washington Avenue, Albany, NY 12206; telephone: (518) 442-4900. Offers therapy on a sliding scale based on income, with low rates for students.
- For intensive outpatient program (IOP) services for eating disorders: HPA/LiveWell located at 260 Washington Avenue Extension, Suite 101, Albany, NY 12203; telephone: (518) 218-1188 [Note: the P.I. in this study (DCW) is on staff at HPA/LiveWell as a clinical psychologist, so is aware of patients seen in the IOP. In this capacity, DCW is legally required to uphold patient confidentiality.]

#### Consent of the participant:

| I have read, or been informed of, the information about thi | s study. I hereby consent to participate in the study. |
|---|---|
| Name: | |
| Signature: | Date: |

# Self-Image Research Study – Informed Consent (C) University at Albany

**Researchers:** D. Catherine Walker, Ph.D., Visiting Assistant Professor of Psychology at Union College and Volunteer Research Associate at University at Albany, State University of New York (Principal Investigator) and Drew A. Anderson, Ph.D., Associate Professor of Psychology at University at Albany, State University of New York, co-Principal Investigator.

**Research Description:** This self image research study aims to test the impact of undergraduate women's response to guided mirror exposure and texts that prompt them to focus on gratitude.

**Human Subject Involvement:** Research participants will be asked to partake in a three-week long program with a one-month and a four month follow-up assessment. All assessment sessions will include answering questions about topics such as mood, self-image, attitudes about the self, self-esteem, and typical self-care behaviors (e.g., eating and physical activity). Each weekly session in the lab will likely last approximately a half hour for the three weeks of participation, as well as for each of the the follow-up assessments.

**Risks and Discomforts of Participation:** We do not anticipate any risk in your participation. It is possible that you may become uncomfortable answering some of the questions. Please note that your participation in this study is completely **voluntary**.

Measures taken to minimize risks and discomfort: Participants will be provided with a list of local and national treatment resources.

**Expected benefits to subjects or to others:** Although we cannot promise you any direct benefit from your participation in this study, the knowledge gained may ultimately benefit other individuals who suffer from body image problems. In addition, you may also gain insight into some aspects of your own self-image and will be introduced to a potentially promising new intervention for self-image.

Confidentiality of records/data: All information obtained in this study is strictly confidential: the researcher promises not to divulge this information, unless disclosure is required by law. Information that you provide (in online questionnaires and via text) will be linked with a unique Participant Identification Number. Your name will only be linked to your Participant Identification Number on a password-protected computer file that can only be accessed by Dr. Walker. Research findings containing group data may be published; however, no personal information or individual questionnaire responses will be published.

**Payment to subject for participation:** If participants choose to withdraw from the study, they will be compensated for the portions of the study that they have completed. The payment schedule is as follows: \$10 for the first week, \$10 for the third week, \$15 for the 1 month follow up assessment, and \$25 for the 4 month follow up assessment - for a **total of \$60** over the course of the study for full participation.

Contact information: If you have any questions about this study, please contact the Principal Investigator: D. Catherine Waker, Ph.D., Licensed Clinical Psychologist and Visiting Assistant Professor of Psychology at Union College, (518)-388-6538, walkerc@union.edu. You will be offered a copy of this form to keep.

**Your rights as a research participant:** Research at Union College involving human participants is carried out under the oversight of the Human Subjects Research Committee (HSRC). This research has been reviewed and approved by the HSRC. If you have any questions about your rights as a human research participant, more information can be found at the Office of Human Research Protections: https://www.hhs.gov/ohrp/

**Voluntary Nature of Participation:** Even after you agree to participate, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise are entitled. You can choose at any time not to answer a question, or not complete a portion of the research for any reason.

Withdrawal of subjects and data retention: Your participation in this project is voluntary. Even after you agree to participate in the research or sign the informed consent document, you may decide to leave the study at any time without penalty or loss of benefits to which you may otherwise have been entitled. I will retain and analyze the information you have provided unless you request that your data be excluded from any analysis and/or destroyed.

Listed below are mental health resources in the even that you have concerns related to or are upset by any of the topics covered in this study.

- For emergency mental health services, call the Albany County Mental Health 24-hour Crisis Hotline at (518) 447-9650 or the Samaritan Hospital 24-Hour Crisis Line at (518) 274-4345.
- The National Eating Disorders Association helpline has a telephone and an online chat support: <a href="https://www.nationaleatingdisorders.org/help-support/contact-helpline">https://www.nationaleatingdisorders.org/help-support/contact-helpline</a>; Confidential helpline, Monday Thursday from 9:00 am 9:00 pm and Friday from 9:00 am 5:00 pm (EST): 1-800-931-2237
- The University at Albany Counseling Center (for UAlbany students) located at 400 Patroon Creek Blvd Suite 104, Albany, NY 12206; email: consultation@albany.edu; telephone: (518) 442-5800.
- The Psychological Services Center located 299 Washington Avenue, Albany, NY 12206; telephone: (518) 442-4900.
- Counseling Care and Services located at 405 Vliet Boulevard, Cohoes, NY 12047; telephone: (518) 237-4263.
- For intensive outpatient program (IOP) services for eating disorders: HPA/LiveWell located at 260 Washington Avenue Extension, Suite 101, Albany, NY 12203; telephone: (518) 218-1188 [Note: the P.I. in this study (DCW) is on staff at HPA/LiveWell as a clinical psychologist, so is aware of patients seen in the IOP. In this capacity, DCW is legally required to uphold patient confidentiality.]

### Consent of the participant:

| ŕ | ŕ | , | • | • | • | • |
|------------|---|---|-------|---|---|---|
| 3.7 | | | | | | |
| Name: | | | | | | |
| Signature: | | | Date: | | | |

I have read, or been informed of, the information about this study. I hereby consent to participate in the study.